CLINICAL TRIAL: NCT00880958
Title: Effects of Supplement Containing Various Probiotics and Fermentation Products on Obesity: a Double-Blind, Randomized Controlled Trial
Brief Title: Effects of Supplement Containing Various Probiotics and Fermentation Products on Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Biostir, Inc. (Industry); MIONA Co., Ltd. (Unknown)
Responsible Party: Fumiko Higashikawa, PhD/Associate professor, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: eki-123
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Mixture of various probiotics and fermentation products
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mixture of various probiotics and fermentation products
  Arms: 1
Dietary Supplement: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of supplement combined various probiotics and fermentation products on body mass index, body fat mass, abdominal circumference, visceral fat mass, intestinal flora, and serum biochemical parameters in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as based on medical history and physical examination
* BMI between 25 and 30 kg/m2
* Willing not to serve as blood donor during the study
* Informed consent signed

Exclusion Criteria:

* Food allergy
* Female subjects who are pregnant or nursing a child
* Participation in any clinical trial up to 90 days before Day 01 of this study
* Renal or hepatic dysfunction
* Heart disease
* Under medication
* Subjects who are taking functional food designed for weight loss or serum lipid reduction

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Body mass index | 16 weeks

SECONDARY OUTCOMES:
Body fat mass | Week -4, Week 0, Week 4, Week 12
Abdominal circumference | Week -4, Week 0, Week 4, Week 12
Visceral fat area by CT scan | Week 0, Week 12
Intestinal flora | Week 0, Week 12
Serum lipid profile | Week -4, Week 0, Week 4, Week 12
Serum adiponectin and leptin levels | Week 0, Week 12
Fasting serum glucose and HbA1c levels | Week -4, Week 0, Week 4, Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan